CLINICAL TRIAL: NCT05140018
Title: Incidence, Course and Outcome of Cellular and Antibody-mediated Rejection in Immunological High-risk Kidney Transplantation, a Prospective Cohort PROCARE2 Study
Brief Title: Incidence, Course and Outcome of ABMR in Kidney Transplantation
Acronym: PROCARE2
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Kidney Foundation (Other); UMC Utrecht (Other); Leiden University Medical Center (Other); Maastricht University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Erasmus Medical Center (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, J.S.F. Sanders, Principal Investigator, University Medical Center Groningen
Other Study IDs: PROCARE2
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Antibody-mediated Rejection; Kidney Transplantation; Immunosuppression
MeSH Terms: interventions — Kidney Transplantation; Immunosuppression Therapy; Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cells (PBMCs) Kidney biopsy material (in case when kidney biopsy is performed in the follow-up) Iliac lymph nodes from 15 selected kidney transplant recipients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kidney Transplant Recipients with an immunological high risk for ABMR: * Kidney transplant recipients ≥18 years old
  * About to receive a post mortal or living donor renal transplant
  * Immunological high risk for rejection
    1. Luminex positive DSAs ; or
    2. Retransplantation with repeated mismatch ; or
    3. Husband to wife donation (after fathering children); or
    4. Offspring to mother donation
  Interventions: Procedure: Kidney Transplantation; Combination Product: Immunosuppression
- Living Kidney Donors: Participants who are about to donate their kidney to a Recipient with a high immunological risk (as described above)
  Interventions: Procedure: Nephrectomy (kidney donation)

INTERVENTIONS:
Procedure: Kidney Transplantation — All participants will receive a kidney transplantation from a living donor or deceased donor
  Groups: Kidney Transplant Recipients with an immunological high risk for ABMR
Combination Product: Immunosuppression — All participants will receive immunosuppresive drugs to prevent rejection of de kidney transplant graft.
  Groups: Kidney Transplant Recipients with an immunological high risk for ABMR
Procedure: Nephrectomy (kidney donation) — All kidney donors will receive a nephrectomy for kidney donation
  Groups: Living Kidney Donors

SUMMARY:
Rationale: Despite improved patient and graft survival in renal transplant recipients, still 20% of the patients reaches end-stage renal disease within 5 years after transplantation. Antibody-mediated rejection (ABMR) is one of the major causes of early graft loss and perhaps even more important of late deterioration of graft function

Objective: Evaluate the occurrence of antibody mediated rejection (ABMR) and mixed ABMR and cellular/ T-cell mediated rejection (TCMR), in patients treated with the currently prevailing immunosuppressive regimens, and relate them to outcome (graft survival, function, proteinuria, histology)

Study design: Clinical cohort study.

Study population: patients of >18 years old, about to receive a post mortal of living donor renal transplant with an immunological high risk for ABMR.

Main study parameters/endpoints: main study endpoints are the occurrence of ABMR, mixed ABMR/TCMR and renal function after 1 year of follow-up.

The main study parameter will be mapping the immune system, including B-cells, (non-)HLA antibodies, interaction between B-cells and T follicular helper cells, and complete immune profiling.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients ≥18 years old
* About to receive a post mortal or living donor renal transplant
* written informed consent (is able to read of understand in Dutch)
* Immunological high risk for rejection

  1. Luminex positive DSAs ; or
  2. Retransplantation with repeated mismatch ; or
  3. Husband to wife donation (after fathering children); or
  4. Offspring to mother donation

Exclusion Criteria:

* No immunological high risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with eind-stage renale disease (ESRD) who are about to receive a kidney transplant from a living or deceased donor, with an elevated immunological risk (higher risk for (antibody-mediated) rejection).
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Antibody-Mediated Rejection (ABMR) | within 12 months after transplantation
  Incidence of Antibody-Mediated Rejection (ABMR) as histopathological diagnosis
Incidence of mixed Antibody-Mediated Rejection / T-Cell Mediated Rejection (ABMR/TCMR) | within 12 months after transplantation
  Incidence of mixed Antibody-Mediated Rejection / T-Cell Mediated Rejection as histopathological diagnosis(ABMR/TCMR) as histopathological diagnosis
Kidney transplant function | at 12 months after transplantation
  as measured by eGFR and proteinuria

SECONDARY OUTCOMES:
Development of Human-Leukocyte Antigen (HLA) antibodies | At 3 and 12 months after transplantation
  As measured by Luminex assay at 3 and 12 months
Development of non-HLA antibodies | At 3 and 12 months after transplantation
  Development of non-HLA antibodies as measured by a cell-based endothelial assay
Kidney transplant survival | At 12 months after transplantation
  Kidney transplant survival in patients experiencing ABMR versus those not experiencing ABMR

CONTACTS AND LOCATIONS:
Overall Officials: Hendrikus Otten, PhD, Study Chair — UMC Utrecht
Locations (6):
- Netherlands (6):
  - Academisch Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Radboud University Hospital, Nijmegen
  - Erasmus MC, Rotterdam
  - UMCU, Utrecht

IPD SHARING:
Plan to Share IPD: No